CLINICAL TRIAL: NCT01919697
Title: An Open-Label Extension (OLE), Long-term Safety and Tolerability Study of Plecanatide in Patients With Chronic Idiopathic Constipation (CIC)
Brief Title: Open-label Extension (OLE) Study of Plecanatide for Chronic Idiopathic Constipation (CIC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP304203-01
Record Dates: First submitted 2013-08-07; First posted 2013-08-09 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Chronic Idiopathic Constipation
Keywords: Plecantaide; Chronic Idiopathic Constipation; Chronic; Idiopathic; Constipation; Synergy; CIC; CIC study; CIC OLE; CIC OLE study; OLE; OLE CIC; OLE CIC3; Open label; Open label study; Long term; Long term study; Extension; Extension study
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Constipation | interventions — plecanatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plecanatide 3.0 mg (Experimental): Plecanatide 3.0 mg, one tablet by mouth daily for 52 weeks
  Interventions: Drug: Plecanatide
- Plecanatide 6.0 mg (Experimental): Plecanatide 6.0 mg, one tablet by mouth daily for 52 weeks
  Interventions: Drug: Plecanatide

INTERVENTIONS:
Drug: Plecanatide

SUMMARY:
This is a multi-center, open-label, 52-week safety and tolerability study of plecanatide in patients with Chronic Idiopathic Constipation (CIC).

DETAILED DESCRIPTION:
This is an open-label extension study of plecanatide in the treatment of patients with CIC who previously completed Synergy Protocols SP304-20210 and SP304203-00 (The CIC3 Study).

The planned duration of each patient's study participation is up to 411 days, including up to 33 days of screening, 8 study visits over 52 weeks of treatment and a follow-up visit 2 weeks after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Patient completed a previous double-blind plecanatide study and was compliant with the study requirements.
* Patient is in good health without unstable acute illness or exacerbation of an unstable chronic illness or chronic disease that may affect study assessments, particularly if there has been a significant change to health status since the previous plecanatide study.

Exclusion Criteria:

* Patient has had major surgery including laparoscopic procedures requiring general anesthesia within 60 days of Day 1.
* Patient has a medical history of hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection.
* Patient has taken a protocol-prohibited drug without the appropriate washout period.

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2370 (Actual)
Dates: Start 2013-08; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Krause, MD, Principal Investigator — ClinSearch, LLC
Locations (171):
- United States (163):
  - Synergy Research Site, Birmingham, Alabama
  - Synergy Research Site, Dothan, Alabama
  - Synergy Research Site, Gulf Shores, Alabama
  - Synergy Research Site, Huntsville, Alabama
  - Synergy Research Site, Chandler, Arizona
  - Synergy Research Site, Phoenix, Arizona
  - Synergy Research Site, Tempe, Arizona
  - Synergy Research Site, Tucson, Arizona
  - Synergy Research Site, Little Rock, Arkansas
  - Synergy Research Site, North Little Rock, Arkansas
  - Synergy Research Site, Anaheim, California
  - Synergy Research Site, Artesia, California
  - Synergy Research Site, Carlsbad, California
  - Synergy Research Site, Cerritos, California
  - Synergy Research Site, Chula Vista, California
  - Synergy Research Site, Corona, California
  - Synergy Research Site, Encinitas, California
  - Synergy Research Site, Fountain Valley, California
  - Synergy Research Site, Fresno, California
  - Synergy Research Site, Hawaiian Gardens, California
  - Synergy Research Site, La Mirada, California
  - Synergy Research Site, Laguna Hills, California
  - Synergy Research Site, Lancaster, California
  - Synergy Research Site, Long Beach, California
  - Synergy Research Site, Los Angeles, California
  - Synergy Research Site, Mission Hills, California
  - Synergy Research Site, North Hollywood, California
  - Synergy Research Site, Orange, California
  - Synergy Research Site, Pasadena, California
  - Synergy Research Site, Sacramento, California
  - Synergy Research Site, San Diego, California
  - Synergy Research Site, Thousand Oaks, California
  - Synergy Research Site, Colorado Springs, Colorado
  - Synergy Research Site, Denver, Colorado
  - Synergy Research Site, Littleton, Colorado
  - Synergy Research Site, Bristol, Connecticut
  - Synergy Research Site, Waterbury, Connecticut
  - Synergy Research Site, Boynton Beach, Florida
  - Synergy Research Site, Brandon, Florida
  - Synergy Research Site, Clearwater, Florida
  - Synergy Research Site, Cutler Bay, Florida
  - Synergy Research Site, DeLand, Florida
  - Synergy Research Site, Fort Lauderdale, Florida
  - Synergy Research Site, Hialeah, Florida
  - Synergy Research Site, Homestead, Florida
  - Synergy Research Site, Jupiter, Florida
  - Synergy Research Site, Lakeland, Florida
  - Synergy Research Site, Miami, Florida
  - Synergy Research Site, Miami Lakes, Florida
  - Synergy Research Site, Miami Springs, Florida
  - Synergy Research Site, Orlando, Florida
  - Synergy Research Site, Pembroke Pines, Florida
  - Synergy Research Site, Port Orange, Florida
  - Synergy Research Site, St. Petersburg, Florida
  - Synergy Research Site, Tamarac, Florida
  - Synergy Research Site, Tampa, Florida
  - Synergy Research Site, West Palm Beach, Florida
  - Synergy Research Site, Athens, Georgia
  - Synergy Research Site, Atlanta, Georgia
  - Synergy Research Site, Decatur, Georgia
  - Synergy Research Site, Oakwood, Georgia
  - Synergy Research Site, Sandy Springs, Georgia
  - Synergy Research Site, Savannah, Georgia
  - Synergy Research Site, Smyrna, Georgia
  - Synergy Research Site, Snellville, Georgia
  - Synergy Research Site, Blackfoot, Idaho
  - Synergy Research Site, Chicago, Illinois
  - Synergy Research Site, Brownsburg, Indiana
  - Synergy Research Site, Clive, Iowa
  - Synergy Research Site, Augusta, Kansas
  - Synergy Research Site, Newton, Kansas
  - Synergy Research Site, Shawnee Mission, Kansas
  - Synergy Research Site, Wichita, Kansas
  - Synergy Research Site, Lexington, Kentucky
  - Synergy Research Site, Owensboro, Kentucky
  - Synergy Research Site, Bastrop, Louisiana
  - Synergy Research Site, Marrero, Louisiana
  - Synergy Research Site, Metairie, Louisiana
  - Synergy Research Site, New Orleans, Louisiana
  - Synergy Research Site, Shreveport, Louisiana
  - Synergy Research Site, Chevy Chase, Maryland
  - Synergy Research Site, Boston, Massachusetts
  - Synergy Research Site, New Bedford, Massachusetts
  - Synergy Research Site, Chesterfield, Michigan
  - Synergy Research Site, Flint, Michigan
  - Synergy Research Site, Rochester, Michigan
  - Synergy Research Site, Saginaw, Michigan
  - Synergy Research Site, Southfield, Michigan
  - Synergy Research Site, Biloxi, Mississippi
  - Synergy Research Site, Jackson, Mississippi
  - Synergy Research Site, St Louis, Missouri
  - Synergy Research Site, Grand Island, Nebraska
  - Synergy Research Site, Omaha, Nebraska
  - Synergy Research Site, Henderson, Nevada
  - Synergy Research Site, Las Vegas, Nevada
  - Synergy Research Site, Reno, Nevada
  - Synergy Research Site, Elizabeth, New Jersey
  - Synergy Research Site, Lodi, New Jersey
  - Synergy Research Site, Marlton, New Jersey
  - Synergy Research Site, Albuquerque, New Mexico
  - Synergy Research Site, Brooklyn, New York
  - Synergy Research Site, Great Neck, New York
  - Synergy Research Site, New York, New York
  - Synergy Research Site, Poughkeepsie, New York
  - Synergy Research Site, Cary, North Carolina
  - Synergy Research Site, Chapel Hill, North Carolina
  - Synergy Research Site, Charlotte, North Carolina
  - Synergy Research Site, Greensboro, North Carolina
  - Synergy Research Site, Kinston, North Carolina
  - Synergy Research Site, Raleigh, North Carolina
  - Synergy Research Site, Wilmington, North Carolina
  - Synergy Research Site, Winston-Salem, North Carolina
  - Synergy Research Site, Fargo, North Dakota
  - Synergy Research Site, Beavercreek, Ohio
  - Synergy Research Site, Centerville, Ohio
  - Synergy Research Site, Cincinnati, Ohio
  - Synergy Research Site, Cleveland, Ohio
  - Synergy Research Site, Huber Heights, Ohio
  - Synergy Research Site, Maumee, Ohio
  - Synergy Research Site, Mentor, Ohio
  - Synergy Research Site, Oakwood, Ohio
  - Synergy Research Site, Stow, Ohio
  - Synergy Research Site, Norman, Oklahoma
  - Synergy Research Site, Oklahoma City, Oklahoma
  - Synergy Research Site, Levittown, Pennsylvania
  - Synergy Research Site, Limerick, Pennsylvania
  - Synergy Research Site, Philadelphia, Pennsylvania
  - Synergy Research Site, Pittsburgh, Pennsylvania
  - Synergy Research Site, Yardley, Pennsylvania
  - Synergy Research Site, Anderson, South Carolina
  - Synergy Research Site, Charleston, South Carolina
  - Synergy Research Site, Columbia, South Carolina
  - Synergy Research Site, Chattanooga, Tennessee
  - Synergy Research Site, Franklin, Tennessee
  - Synergy Research Site, Jackson, Tennessee
  - Synergy Research Site, Knoxville, Tennessee
  - Synergy Research Site, Memphis, Tennessee
  - Synergy Research Site, Nashville, Tennessee
  - Synergy Research Site, New Tazewell, Tennessee
  - Synergy Research Site, Arlington, Texas
  - Synergy Research Site, Austin, Texas
  - Synergy Research Site, Channelview, Texas
  - Synergy Research Site, Dallas, Texas
  - Synergy Research Site, Houston, Texas
  - Synergy Research Site, Humble, Texas
  - Synergy Research Site, Katy, Texas
  - Synergy Research Site, Plano, Texas
  - Synergy Research Site, San Antonio, Texas
  - Synergy Research Site, Sugar Land, Texas
  - Synergy Research Site, Logan, Utah
  - Synergy Research Site, Salt Lake City, Utah
  - Synergy Research Site, St. George, Utah
  - Synergy Research Site, West Jordan, Utah
  - Synergy Research Site, Christiansburg, Virginia
  - Synergy Research Site, Henrico, Virginia
  - Synergy Research Site, Lynchburg, Virginia
  - Synergy Research Site, Newport News, Virginia
  - Synergy Research Site, Norfolk, Virginia
  - Synergy Research Site, Richmond, Virginia
  - Synergy Research Site, Richland, Washington
  - Synergy Research Site, Seattle, Washington
  - Synergy Research Site, Tacoma, Washington
  - Synergy Research Site, Wauwatosa, Wisconsin
- Canada (8):
  - Synergy Research Site, Kelowna, British Columbia
  - Synergy Research Site, Bridgewater, Nova Scotia
  - Synergy Research Site, Cambridge, Ontario
  - Synergy Research Site, Greater Sudbury, Ontario
  - Synergy Research Site, Toronto, Ontario
  - Synergy Research Site, Mirabel, Quebec
  - Synergy Research Site, Pointe-Claire, Quebec
  - Synergy Research Site, Saint Romuald, Quebec

REFERENCES:
- [Derived] Barish CF, Griffin P. Safety and tolerability of plecanatide in patients with chronic idiopathic constipation: long-term evidence from an open-label study. Curr Med Res Opin. 2018 Apr;34(4):751-755. doi: 10.1080/03007995.2018.1430024. Epub 2018 Feb 2. PMID 29343131

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with CIC who completed the double-blind phase 2b (NCT01429987) study, or phase 3 (NCT01982240 or NCT0222471) studies or who screen-failed for the phase 3 studies due solely to pre-treatment diary compliance and met all of the inclusion criteria and none of the exclusion criteria enrolled into this open-label study.
Pre-assignment Details: A total of 2370 enrolled patients who had received at least one dose of the study drug constituted the Safety Population.
Groups:
- Plecanatide 3 mg: Plecanatide 3 mg, one tablet by mouth daily for up to 72 weeks
- Plecantide 6 mg: Plecanatide 6 mg, one tablet by mouth daily for up to 72 weeks
Period: Overall Study
Arm/Group | Plecanatide 3 mg | Plecantide 6 mg
Started | 224 | 2146
Completed | 171 | 1761
Not Completed | 53 | 385

BASELINE CHARACTERISTICS:
Population: A total of 2321 patients were based on the Safety Population (2370) excluding all duplicate patients except identified as "Index" patients. "Index" was duplicate patients appeared the first time in the enrollment.
Groups:
- Plecanatide 6 mg: Plecanatide 6 mg, one tablet by mouth daily for up to 72 weeks
- Total: Total of all reporting groups
Arm/Group | Plecanatide 3 mg | Plecanatide 6 mg | Total
Number analyzed (Participants) | 224 | 2097 | 2321
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (11.78) | 46.8 (14.03) | 47.0 (13.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 1687 | 1877
  Male | 34 | 410 | 444

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With at Least One Treatment-Emergent Adverse Event (TEAE)
Description: All clinically significant findings upon Physical Examinations of the Safety Population during the treatment period were reported as TEAEs. Safety was evaluated based on number of patients who experienced at least one TEAE.
Time Frame: From first dose up to 72 weeks
Population: The Safety Population consisted of all enrolled patients who had received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Plecanatide 3 mg: Plecanatide 3 mg, one tablet by mouth daily for 72 weeks
- Plecantide 6 mg: Plecanatide 6 mg, one tablet by mouth daily for 72 weeks
Arm/Group | Plecanatide 3 mg | Plecantide 6 mg
Number analyzed (Participants) | 224 | 2146
Participants | 123 | 620

2. Primary Outcome: Number of Patients With at Least One Treatment-Emergent Adverse Event (TEAE) Leading to Discontinuation of Plecanatide
Description: Tolerability was evaluated based on number of patients who experienced at least one TEAE leading to discontinuation of the study drug
Time Frame: From first dose up to 72 weeks
Population: The Safety Population consisted of all enrolled patients who had at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Plecanatide 3 mg | Plecantide 6 mg
Number analyzed (Participants) | 224 | 2146
Participants | 14 | 111

3. Primary Outcome: Summary of Vital Signs at >Day 364 - Blood Pressure (Systolic and Diastolic; mmHg)
Description: The vital signs included in the assessments were blood pressure (systolic and diastolic; mmHg), heart rate (beats per minute), body temperature (°C) and respiration rate (breaths per minute).
Time Frame: From first dose up to 72 weeks
Population: This population (2378 patients) consisted of the Safety Population and the re-enrolled patients who previously participated and completed this open-label study.
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: Readings
Arm/Group | Plecanatide 3 mg | Plecantide 6 mg
Number analyzed (Participants) | 224 | 2146
Number analyzed (Readings) | 224 | 2154
mmHg
  Systolic Blood Pressure | 121 (13.40) | 122.9 (14.11)
  Diastolic Blood Pressure | 75.7 (9.19) | 76.5 (8.47)

4. Primary Outcome: Summary of Vital Signs at >Day 364 - Heart Rate (Beats Per Minute)
Description: as for outcome 3
Time Frame: From first dose up to 72 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beats per minute
Units Other Than Participants: Readings
Arm/Group | Plecanatide 3 mg | Plecantide 6 mg
Number analyzed (Participants) | 224 | 2146
Number analyzed (Readings) | 224 | 2154
beats per minute | 71.2 (10.03) | 71.9 (9.30)

5. Primary Outcome: Summary of Vital Signs at >Day 364 - Body Temperature (°C)
Description: as for outcome 3
Time Frame: From first dose up to 72 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: °C
Units Other Than Participants: Readings
Arm/Group | Plecanatide 3 mg | Plecantide 6 mg
Number analyzed (Participants) | 224 | 2146
Number analyzed (Readings) | 224 | 2154
°C | 36.62 (0.329) | 36.59 (0.378)

6. Primary Outcome: Summary of Vital Signs at >Day 364 - Respiration Rate (Breaths Per Minute)
Description: as for outcome 3
Time Frame: From first dose up to 72 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: breaths per minute
Units Other Than Participants: Readings
Arm/Group | Plecanatide 3 mg | Plecantide 6 mg
Number analyzed (Participants) | 224 | 2146
Number analyzed (Readings) | 224 | 2154
breaths per minute | 15.7 (2.03) | 16.0 (2.31)

7. Primary Outcome: Summary of ECG Results Shift From Baseline at > Day 364
Description: Baseline was defined as the last non-missing value collected prior to first dose of study drug)
Time Frame: From first dose up to 72 weeks
Population: as for outcome 3
Measure: Number; unit: participants
Units Other Than Participants: Readings
Arm/Group | Plecanatide 3 mg | Plecantide 6 mg
Number analyzed (Participants) | 224 | 2146
Number analyzed (Readings) | 224 | 2154
participants
  Change from Normal to Abnormal | 27 | 42
  Change from Adnormal to Normal | 15 | 44

8. Primary Outcome: Summary of Treatment-Emergent Laboratory Abnormalities With At Least a 1-grade Shift From Baseline
Description: Baseline was defined as the last non-missing value collected prior to first dose of study drug within a given entry into the study. The Common Terminology Criteria for Adverse Events (CTCAE), Grades 1 through 5 were used for descriptions of severity for each Adverse Event (AE): Grade 1 - Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; Grade 2 - Moderate; minimal, local or noninvasive intervention indicated; limiting age appropriate instrumental Activities of Daily Living (ADL); Grade 3 - Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL; Grade 4 - Life-threatening consequences; urgent intervention indicated; Grade 5 - Death related to AE.
Time Frame: From first dose up to 72 weeks
Population: as for outcome 3
Measure: Number; unit: participants
Units Other Than Participants: Readings
Arm/Group | Plecanatide 3 mg | Plecantide 6 mg
Number analyzed (Participants) | 224 | 2146
Number analyzed (Readings) | 224 | 2154
participants | 192 | 1498

9. Secondary Outcome: Summary of Patient Patient Global Assessment (PGA) for Constipation Severity at > Day 364
Description: Constipation severity was measured using a 5-point score: 1=None, 2=Mild, 3=Moderate, 4=Severe, 5=Very severe Baseline was defined as the last non-missing value collected prior to first dose of study drug within a given entry into the study.
Time Frame: Form first dose up to 72 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Readings
Arm/Group | Plecanatide 3 mg | Plecantide 6 mg
Number analyzed (Participants) | 224 | 2146
Number analyzed (Readings) | 224 | 2154
score on a scale | 1.8 (0.94) | 1.7 (0.89)

10. Secondary Outcome: Summary of Patient Global Assessment (PGA) for Constipation - Change From Baseline to > Day 364
Description: Change of Constipation measured using a 7-point score: 1=Very Much Improved, 2=Much Improved, 3=Minimally Improved, 4=No change, 5=Minimally Worse, 6=Much Worse, 7=Very Much Worse Baseline is defined as the last non-missing value collected prior to first dose of study drug within a given entry into the study.
Time Frame: From first dose up to 72 weeks
Population: All enrolled patients who had at least one dose of the study drug and had at least one post-baseline Patient Global Assessment (PGA) were included in this population. A total of 2378 patients including the re-enrolled patients who previously participated and completed this open-label study was used for assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Readings
Arm/Group | Plecanatide 3 mg | Plecantide 6 mg
Number analyzed (Participants) | 224 | 2146
Number analyzed (Readings) | 224 | 2154
score on a scale | 1.8 (0.94) | 1.7 (0.89)

11. Secondary Outcome: Summary of Patient Global Assessment (PGA) for Treatment Satisfaction at > Day 364
Description: Baseline was defined as the last non-missing value collected prior to first dose of study drug within a given entry into the study. Treatment Satisfaction was measured using a 5-point score: 1=Not At All Satisfied, 2=A Little Satisfied, 3=Moderately Satisfied, 4=Quite Satisfied, 5=Very Satisfied.
Time Frame: From first dose up to 72 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Readings
Arm/Group | Plecanatide 3 mg | Plecantide 6 mg
Number analyzed (Participants) | 224 | 2146
Number analyzed (Readings) | 224 | 2154
score on a scale | 4.1 (1.13) | 4.2 (1.02)

12. Secondary Outcome: Summary of Patient Global Assessment (PGA) for Treatment Continuation at End of Treatment
Description: Treatment continuation was measured using 5-point score: 1=Not At All Likely, 2=A Little Likely, 3=Moderately Likely, 4=Quite Likely, 5=Very Likely
Time Frame: From first dose up to 72 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Readings
Arm/Group | Plecanatide 3 mg | Plecantide 6 mg
Number analyzed (Participants) | 224 | 2146
Number analyzed (Readings) | 224 | 2154
score on a scale | 4.1 (1.22) | 4.1 (1.16)

ADVERSE EVENTS:
Description: All enrolled patients (2370) who received at least one dose of study drug was included in the risk analysis. There was one death, unrelated to study drug, reported in this study; the patient died from a myocardial infarction (MI) that was related to a cocaine-induced coronary vasopasm.
Groups:
- Plecanatide 6 mg: Plecanatide 6 mg, one tablet by mouth daily for 72 weeks
Arm/Group | Plecanatide 3 mg | Plecanatide 6 mg
All-Cause Mortality (participants affected / at risk) | 0/224 | 1/2146
Serious Adverse Events (participants affected / at risk) | 8/224 | 32/2146
Other Adverse Events (participants affected / at risk) | 32/224 | 188/2146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plecanatide 3 mg (N=224) | Plecanatide 6 mg (N=2146)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 7 (7)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Aspartate aminotransferase abnormal (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram change (Investigations) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plecanatide 3 mg (N=224) | Plecanatide 6 mg (N=2146)
Diarrhoea (Gastrointestinal disorders) | 19 (24) | 150 (159)
Urinary tract infection (Infections and infestations) | 13 (15) | 38 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes